CLINICAL TRIAL: NCT02351635
Title: Clinical Study of the BÜHLMANN fCAL™ ELISA as an Aid in the Differentiation of Inflammatory Bowel Disease From Irritable Bowel Syndrome
Brief Title: BÜHLMANN fCAL™ ELISA - Aid in Differentiation of IBD From IBS
Status: Completed | Type: Observational
Sponsor: Bühlmann Laboratories AG (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Other Study IDs: ALP Cal01
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Inflammatory Bowel Disease; Irritable Bowel Syndrome
Keywords: Calprotectin; Diagnosis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stool samples collected before start of specific medication
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- IBD: Adult subjects with inflammatory bowel disease, confirmed by endoscopy and histologic support. Fecal calprotectin Level.
  Interventions: Other: fecal calprotectin level
- IBS: Adult subjects with Irritable Bowel Syndrome meeting the Rome III criteria. Fecal calprotectin Level.
  Interventions: Other: fecal calprotectin level
- other GI disorders: Adult subjects with gastrointestinal disorders other than IBD or IBS. Fecal calprotectin Level.
  Interventions: Other: fecal calprotectin level
- pediatric: Pediatric patients (2-21 y) diagnosed with IBD, IBS, or other gastrointestinal disorders. Fecal calprotectin Level.
  Interventions: Other: fecal calprotectin level
- healthy controls: Normal adult subjects with no abdominal complaints. Fecal calprotectin Level.
  Interventions: Other: fecal calprotectin level

INTERVENTIONS:
Other: fecal calprotectin level — Stool sample collected by the subject, sent study laboratories where fecal calprotectin levels are quantified.

SUMMARY:
The purpose of this study is to confirm the sensitivity and specificity of the BÜHLMANN fCAL™ ELISA as an aid in diagnosis to differentiate between Inflammatory Bowel Disease (IBD; Crohn's Disease (CD), Ulcerative Colitis (UC), or indeterminate colitis) and Irritable Bowel Syndrome (IBS).

To estimate the predictive value of a positive test (positive predictive value (PPV)) and the predictive value of a negative test (Negative Predictive Value (NPV)) using the proposed test outcomes for BÜHLMANN Calprotectin Test results when used in patients referred for diagnostic evaluation with signs and symptoms suggestive of either IBS or IBD.

To confirm the inter-laboratory consistency of test results for the BÜHLMANN fCAL™ ELISA.

To provide exploratory observations of test results in patients between the age of 2 and 21 years.

To provide a sample set from normal subjects with no symptoms or signs of gastrointestinal disease for use in Expected Value Testing.

ELIGIBILITY:
Inclusion Criteria:

1. Adults or pediatric patients evaluated by a gastroenterological service for investigation of possible inflammatory intestinal disease or IBS. Patients are referred for sub-specialty evaluation of symptoms such as abdominal pain, diarrhea, altered appetite, weight loss, or anemia.

   * IBD: Eligible subjects will be analyzed as patients with IBD after a confirmed diagnosis of Inflammatory Bowel Disease (CD, UC, or Indeterminate Colitis), based on endoscopy and confirmed by histology of biopsies taken during endoscopy.
   * IBS: Eligible candidate subjects can also include patients who are self-referred with the relevant constellation of complaints. Eligible subjects will be enrolled after having a diagnosis of IBS based on the Rome III criteria confirmed by negative endoscopy including the colon and terminal ileum.
   * other GI Disorders: Eligible subjects will be enrolled after having a diagnosis of a gastrointestinal disorder other than IBD or IBS, confirmed by endoscopy results and other appropriate diagnostic studies.
   * Healthy Controls: Adults (≥22) with no abdominal complaints and no history of IBS, IBD or other chronic intestinal disorder, confirmed by medical history and physical examination at enrolment.
2. Individuals of either gender, ≥22 years of age (adult samples) or 2 to -21 years of age (pediatric samples).
3. IBD patients whose diagnostic endoscopy occurred within the previous month.
4. Individuals able to understand the study and the tasks required, and who sign the Informed Consent Form (adult subjects; ICF) or whose parent/guardian provides consent (ICF) and, if age 7-to-18 years of age, who provide assent (pediatric subjects).

Exclusion Criteria:

1. Individuals unable or unwilling to provide a stool specimen.
2. Individuals with known intestinal cancer, intestinal infection, upper gastrointestinal disease
3. Individuals receiving chemotherapy or systemic immunosuppressive drugs.
4. Individuals who have taken, within the previous 2 weeks, protein pump inhibitors or H2-receptor antagonists.
5. Individuals with previously diagnosed Inflammatory Bowel Disease managed with immunomodulators, 5-ASA (5-aminosalicylic acid) or biologic therapies or who have undergone a surgical resection or diversion procedure.
6. Individuals who have taken NSAIDs (nonsteroidal anti-inflammatory drugs), including aspirin, on 7 or more days during the 2 weeks before providing the sample.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 adult subjects with Inflammatory Bowel Disease or Irritable Bowel Syndrome each have provided a stool sample. In addition, 50 pediatric subjects, age 2 years to 21 years, 25 subjects in each diagnostic group (IBD, IBS) will be enrolled. Recruitment of 120 normal subjects who will provide samples.
Sampling Method: Probability Sample
Enrollment: 478 (Actual)
Dates: Start 2015-01; Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Clinical value of in vitro diagnostic (IVD) device | End of Study
  Sensitivity, specificity; Positive predictive value (PPV), negative predictive value (NPV) and likelihood ratios (positive and negative)

SECONDARY OUTCOMES:
normal Calprotectin values | End of Study
  Calprotectin values from normal healthy donors will be calculated
Clinical value of IVD device in pediatric population | End of Study
  Results of the pediatric population will be used as preliminary and exploratory evidence that calprotectin test can be used in this population

OTHER OUTCOMES:
IVD Device performance | 2 months
  The inter-laboratory precision of the device will be investigated across the study laboratories involved.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Gorman, Study Director — ICON Clincal Research
Locations (7):
- United States (7):
  - Stanford Center for Clinical & Translational Research & Education, Palo Alto, California
  - Gastro Health, Miami, Florida
  - Gastroenterology Assocaites of Central Georgia, Macon, Georgia
  - Carle Foundation, Center for Digestive and Liver Disease, Urbana, Illinois
  - Beth israel Deaconess Medical Center, Boston, Massachusetts
  - Great Lakes Gastroenterology Research, LLC., Mentor, Ohio
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manz M, Burri E, Rothen C, Tchanguizi N, Niederberger C, Rossi L, Beglinger C, Lehmann FS. Value of fecal calprotectin in the evaluation of patients with abdominal discomfort: an observational study. BMC Gastroenterol. 2012 Jan 10;12:5. doi: 10.1186/1471-230X-12-5. PMID 22233279
- [Background] Occhipinti K, Smith JW. Irritable bowel syndrome: a review and update. Clin Colon Rectal Surg. 2012 Mar;25(1):46-52. doi: 10.1055/s-0032-1301759. PMID 23449495
- [Background] Kappelman MD, Moore KR, Allen JK, Cook SF. Recent trends in the prevalence of Crohn's disease and ulcerative colitis in a commercially insured US population. Dig Dis Sci. 2013 Feb;58(2):519-25. doi: 10.1007/s10620-012-2371-5. Epub 2012 Aug 29. PMID 22926499
- [Background] Burri E, Beglinger C. Faecal calprotectin -- a useful tool in the management of inflammatory bowel disease. Swiss Med Wkly. 2012 Apr 5;142:w13557. doi: 10.4414/smw.2012.13557. eCollection 2012. PMID 22481443
- [Background] van Rheenen PF, Van de Vijver E, Fidler V. Faecal calprotectin for screening of patients with suspected inflammatory bowel disease: diagnostic meta-analysis. BMJ. 2010 Jul 15;341:c3369. doi: 10.1136/bmj.c3369. PMID 20634346